CLINICAL TRIAL: NCT04764123
Title: To Investigate Whether Remnants of the "Ring Tissues" Constitute the Substrate of the Circuit of Atrioventricular Nodal Reentrant Tachycardia
Brief Title: Typical and Atypical AVNRT High-resolution Mapping
Acronym: AVNRTmap
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cardiovascular Research Society, Greece (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Dr D Katritsis, Director, Cardiovascular Research Society, Greece
Other Study IDs: 2021
Record Dates: First submitted 2021-01-23; First posted 2021-02-21 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Tachycardia, Atrioventricular Nodal Reentry
Keywords: Atrioventricular; Nodal Reentry; Tachycardia
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry; Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AVNRT Cohort: Patients admitted for electrophysiological study and ablation due to AVNRT tachycardia.
  During the study and before the ablation high density electroanatomical mapping will be performed.
  Interventions: Diagnostic Test: AVNRT mapping

INTERVENTIONS:
Diagnostic Test: AVNRT mapping — AV annuli mapping during AVNRT
  Other Names: Electroanatomic mapping

SUMMARY:
This study is aimed at :

1. Identifying the exact location of the circuit of typical and atypical AVNRT by applying high-resolution electroanatomic mapping.
2. Investigating the possibility that the recently described "ring tissues" participate in the AVNRT circuit.

DETAILED DESCRIPTION:
Background The exact circuit of atrioventricular nodal reentrant tachycardia still remains unknown despite advances in high-density mapping, tissue histochemistry, and connexin genotyping. Theoretical calculations have derived a range of 0.8 to 5.2 cm for the length of the slow pathway, whereas that of the fast pathway should be within the range of 2.4 to 11.2 cm. Recent histology data also indicate that the distance of the right inferior extension of the atrioventricular node within the tricuspid vestibule, as judged histologically, and as measured from the site of penetration of the conduction axis in 31 hearts, is 8.2±2.4 mm, with a range from 5.2 to 13.6 mm. These results are compatible with theoretical calculations of the slow pathway previously performed by the investigators. On 3-dimensional reconstructed fluoroscopic images, the average distance between the compact AV node and the ablating electrode in cases of successful AVNRT ablation, however, is 17.2±1.6 to 17.8±0.9 mm. This clearly suggests that successful ablation interrupts the AVNRT circuit at a point beyond the identifiable right posterior extension, and at a consistent area on the the septal isthmus between the CS ostium and the TV. This site is beyond the histologically identifiable inferior extensions of the node.

There is additional evidence in animal studies that the right inferior extension continues within the vestibule of the tricuspid valve as "ring tissue", ie a remnant of the primary ring, while the left atrial vestibule is derived from the initial atrioventricular canal of the developing heart, which is itself known to be slow conducting but cannot be distinguished histologically from the left atrial myocardium. In the human heart, the primary ring extends through the atrioventricular node, and includes the bundle of His, which is rapidly conducting.

Hypothesis The investigators hypothesized that, in humans, the extent of ring tissues varies in such a way that some subjects are susceptible to atrioventricular nodal re-entry, whereas others are not. Thus, the entirety of the tricuspid vestibule, or even part of the mitral vestibule, are parts of the re-entry circuit, at least in some atypical forms with prolonged His-atrial intervals. The circumference of the right atrioventricular orifice has been measured at between 9 and 11 centimeters in patients aged less than 65 years, whereas that of the mitral orifice is from 7 to 9 centimeters. The possibility of the vestibules being involved in the circuit, therefore, cannot theoretically be excluded. Recently, high-density mapping of the re-entry circuit has provided valuable insights into the electrophysiologic patterns of this arrhythmia, identifying the circuit in the vicinity of the nodal area. All these mapping studies, however, were conducted in patients with typical AVNRT. In this setting, the remnants of the ring tissues might be short enough as not to allow proper discrimination of the circuit limbs. The investigators propose to apply high-resolution electroanatomic mapping in patients with both typical atypical AVNRT in which the circuit may contain longer circuit components. Mapping should be focused on both the septal area and the tricuspid, and, if feasible, the mitral ring.

Aims of the Study

This study, therefore, is aimed at :

1. Identifying the exact location of the circuit of typical and atypical AVNRT by applying high-resolution electroanatomic mapping.
2. Investigating the possibility that the recently described "ring tissues" participate in the AVNRT circuit.

Methods Clinical Studies Patients Patients with typical and atypical AVNRT will be recruited following informed consent. The investigators anticipate to study 30 patients with typical, and 10 patients with atypical AVNRT within the next two years.

Definitions AVNRT is diagnosed by fulfillment of established criteria during detailed atrial and ventricular pacing maneuvers. Typical (slow-fast) AVNRT is defined by an atrial-His/His-atrial ratio (AH/HA) >1, and HA interval ≤70 ms. Atypical AVNRT is defined by delayed retrograde atrial activation with HA>70 ms.

Mapping Electroanatomic mapping will be performed with CARTO, Rhythmia or Ensite programs at the operator's discretion. High-resolution mapping of the atrial vestibules is inherently difficult in this setting, nonetheless, because of the problems in separating a large ventricular electrogram from the atrial tracing. During atrioventricular nodal reentry, all these areas should show a fused signal consisting of nodal activation. Any mapping system will struggle to annotate the fused signal appropriately in the window and during tachycardia. It may also preferentially annotate the His bundle electrogram because of its high frequency (dv/dt). The implication of this error is that a site annotated as representing the earliest atrial activity may be representing activity in the His bundle. Conversely, a site marked as late may, in fact, be early, being obscured by far field ventricular activity. These limitations may also apply to animal models using micro-electrode mapping. To overcome this problem, pacing maneuvers with ventricular extrastimuli are used to differentiate atrial from ventricular electrogram components where activation appeared to be superimposed owing to simultaneous local activation. In addition, the investigators will exclude points that result in discrepant activation relative to the surrounding isochronal information due to the movement of the CS reference catheter. Activation points from ectopic beats will be excluded manually. The voltage map will be automatically acquired according to the same criteria. After automated mapping, an offline retrospective analysis will be performed by 2 independent observers, in order to manually over-read the sites of earliest atrial activation, at an override activation strength of 100 mV in cases in which (1) the earliest activation on automated mapping appeared diffuse or (2) automated annotation tagged the local ventricular component at the annulus. The His-bundle signal is generally automatically annotated by the system.

Entrainment Entrainment of AVNRT is feasible at sites close to the nodal extensions. Attempts will be made to entrain the tachycardia from various points on the TV annulus in order to investigate potential participation of the right-sided ring tissue into circuit.

Catheter ablation Being on the operation discretion, before conventional catheter ablation of the slow pathway, at least two 30 sec lesions will be delivered on the TV annulus near the isthmus, if this feasible. Interruption of the tachycardia or evoked junctional beats will be sought. Conventional catheter ablation of the slow pathway will be performed as previously described.

Histology Studies Databases from human hearts specimens will be examined and tissue-characterized in an attempt to identify the presence and extent of "ring tissues" in the human myocardium.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atypical or typical AVNRT
* Patients able to provide informed consent

Exclusion Criteria:

* Age <16 or >75 years
* Known heart failure
* Severe comorbidities with estimated life expectancy < 6 months

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with typical or atypical AVNRT admitted for electrophysiological study and ablation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Participation of ring tissues in the AVNRT Circuit | 2 years
  Tachycardia entrainment by pacing at the anatomical ring tissue site or tachycardia termination with successful ablation at the ring tissue site

SECONDARY OUTCOMES:
Fast and slow pathway activation time in the circuit of AVNRT. | 2 years
  TIme in ms required for fast and slow pathway activation during tachycardia.